CLINICAL TRIAL: NCT01895894
Title: A Prospective, Randomized, Open-label Study Evaluating the Efficacy of Mycophenolate Mofetil in the Prevention of Relapse of Steroid Dependent Nephrotic Syndrome in Children
Brief Title: Mycophenolate Mofetil in Pediatric Steroid Dependent Nephrotic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Hee Gyung Kang, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMF2013
Record Dates: First submitted 2013-07-07; First posted 2013-07-11 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Nephrotic Syndrome
Keywords: Mycophenolate mofetil; Immunosuppressive Agents; Nephrosis
MeSH Terms: conditions — Nephrotic Syndrome; Nephrosis | interventions — Mycophenolic Acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolate mofetil (Experimental)
  Interventions: Drug: Mycophenolate mofetil
- Control (No Intervention)

INTERVENTIONS:
Drug: Mycophenolate mofetil — Mycophenolate mofetil 20~30mg/kg/day PO until nephrotic syndrome relapse (max. 1 year)
  Other Names: Myrept capsule/tablet
  Arms: Mycophenolate mofetil

SUMMARY:
Idiopathic nephrotic syndrome is generally responsive to steroid therapy, but some patients need other immunosuppressants to reduce steroid dependency. The long-term use should be restricted due to adverse effects of cyclosporine, such as hypertension and nephrotoxicity.

Mycophenolate mofetil for steroid-dependent nephrotic syndrome has been reported to have similar efficacy and fewer undesirable effects to other drugs in mainly observational studies. To determine the efficacy of mycophenolate mofetil in the management of steroid-dependent nephrotic syndrome, the investigators designed this prospective randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Steroid-dependent patients who had been on calcineurin inhibitors continuously for more than 1 year
* in complete remission

Exclusion Criteria:

* Hereditary or secondary nephrotic syndrome
* Estimated glomerular filtration rate (GFR) < 60 mg/min/1.73 m^2
* Body weight <16 kg
* leukocytopenia (absolute neutrophil count < 2000/mm^3) or anemia(Hct < 25%)
* Severe gastrointestinal disease
* chronic or acute active infection (e.g. hepatitis B,C, herpes, varicella zoster)
* prior live vaccine inoculation within 6 weeks (from the study enrollment)
* GOT/GPT elevation or hyperbilirubinemia
* malignant disease
* Pregnant or Breast feeding
* Previous history of mycophenolate mofetil use
* Participation to other therapeutic trial within recent 3 months
* Deficiency of the enzyme hypoxanthine-guanine phosphoribosyltransferase

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
relapse free time | 1 year

SECONDARY OUTCOMES:
adverse effect | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hee Gyung Aurea Kang, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526